CLINICAL TRIAL: NCT00364104
Title: Randomized Field Intervention Trial of H. Pylori Eradication to Reduce Iron Deficiency Among Children in El Paso, Texas
Brief Title: Helicobacter Pylori Eradication Trial to Reduce Iron Deficiency in Children
Acronym: HEIDC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Texas Tech University (Other); University of Texas (Other); Baylor College of Medicine (Other); University of North Texas Health Science Center (Other)
Responsible Party: Victor M. Cardenas, MD, MPH, PhD, Associate Professor, UT Houston HSC School of Public Health El Paso Regional Campus
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: HSC-SPH-06-0374
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Iron Deficiency
Keywords: Iron deficiency; Helicobacter infection; Epidemiology
MeSH Terms: conditions — Iron Deficiencies; Helicobacter Infections | interventions — Iron-Dextran Complex; ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Experimental): A 10-day course of Hp infection sequential eradication therapy plus 6-weeks of iron supplementation
  Interventions: Drug: Quadruple sequential Helicobacter pylori eradication + iron sulfate
- B (Experimental): The 10-day course of Hp infection sequential eradication therapy only plus 6-weeks of matching placebo of iron supplementation
  Interventions: Drug: Quadruple sequential Helicobacter pylori eradication therapy
- C (Experimental): 6-weeks of iron supplementation only plus 10-days of matching placebo of Hp infection eradication therapy
  Interventions: Drug: Ferrous sulfate
- D (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quadruple sequential Helicobacter pylori eradication + iron sulfate — A 10-day course of Hp infection sequential eradication therapy plus 6-weeks of iron supplementation
  Arms: A
Drug: Quadruple sequential Helicobacter pylori eradication therapy — A 10-day course of Hp infection sequential eradication therapy only plus 6-weeks of matching placebo of iron supplementation
  Arms: B
Drug: Ferrous sulfate — 6-weeks of iron supplementation only plus 10-days matching placebo of Hp infection eradication therapy
  Arms: C
Drug: Placebo — Placebo only (10-days of matching placebo of Hp eradication therapy and 6-weeks of matching iron supplementation).
  Arms: D

SUMMARY:
The investigators hypothesize that the Helicobacter pylori bacterium decreases iron from the stomach and that this effect of the infection can be identified among persons with iron deficiency as well as among persons with normal iron stores. The aim of this study is to determine whether Helicobacter pylori eradication in children is followed by an increase in markers of iron stores after six to twelve months of treatment.

DETAILED DESCRIPTION:
For the last 12 years, scientific evidence has mounted linking Helicobacter pylori infection with iron deficiency and iron deficiency anemia. Reports from around the world on several cases of iron deficiency anemia refractory to iron supplementation among children infected with Helicobacter pylori, most without evident ulcers, clearly indicate that such cases have been cured of their anemia after receiving a course of Helicobacter pylori eradication therapy. Several studies based on national surveys, including one on the U.S. National Health and Nutrition Examination Survey data and conducted by the authors of this proposal, have found an association between Helicobacter pylori infection and the levels of iron stores. However, these studies fail to demonstrate that anemia follows Helicobacter pylori infection. Moreover, most previous research has been conducted outside of the contiguous U.S. and has not included young children, one of the high-risk populations for iron deficiency and iron deficiency anemia. Data on this age-group is most needed to develop sound public health interventions.

We propose to conduct such a study among children living in El Paso, Texas, a city located on the U.S.-Mexico border. A series of studies have been conducted in that city by the authors of this proposal, including a National Institutes of Health sponsored study aiming to describe the natural history of Helicobacter pylori infection in children from birth to age seven years (84 months). We hypothesize that the Helicobacter pylori bacterium decreases iron from the stomach and that this effect of the infection can be identified among persons with iron deficiency as well as among persons with normal iron stores. Currently, the clinical management of the most extreme form of iron deficiency, that is iron deficiency anemia, relies only on supplemental iron therapy. For ethical reasons, our study will identify children with anemia from the study, and will assign them to one of the arms receiving iron supplementation. Our study will determine whether a combination of iron supplementation and sequential Helicobacter pylori eradication therapy yields higher increases of iron stores than each of these treatments alone. To summarize, our main hypothesis is that Helicobacter pylori infection is associated with iron deficiency such that Helicobacter pylori eradication would result in an increase in the levels of:

1. serum ferritin,
2. transferrin saturation, and
3. hemoglobin.

To test these hypotheses we will randomly assign 125 Helicobacter pylori-infected children (3 to 10 years of age) into each of the following four groups: Helicobacter pylori eradication treatment, iron supplementation, Helicobacter pylori eradication plus iron supplementation, or placebo. We plan to recruit infected children through a household survey in El Paso, screen their Helicobacter pylori infection status by a stool test, and invite their parents to undergo a confirmatory breath test. Infected children randomly allocated to those four arms of the study will be followed closely during the 6 weeks they are taking the study medication to record any adverse event, followed by a visit at 45 days after treatment to tell whether or not those receiving the medication had their infection eradicated, between 6 and 12 months for hematological evaluation to compare with the baseline levels of iron stores.

ELIGIBILITY:
Inclusion Criteria:

* Children 3-10 years of age
* Helicobacter pylori infected, asymptomatic
* Healthy otherwise
* Parents provided consent/assenting children 7-10 years of age

Exclusion Criteria:

* Parental consent or child assent not obtained
* History of antibiotic-related allergic episodes
* Children with a history of allergy, asthma, hay fever or urticaria
* Phenylketonurics
* Abnormal renal and hepatic functions as evaluated through albumin, bilirubin, AST (or SGOT), ALT (or SGPT), alkaline phosphatase and GGT-P
* History of peptic ulcer
* History of recent (< 1 month) severe disease
* History of recent (< 1 month) use of antibiotics, antacids, H2 receptor antagonists, proton pump inhibitors and remedies containing bismuth
* Parents uncertain about staying in El Paso for the next year

Ages: 36 Months to 120 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Percent change of serum ferritin | between 6 and 12 months
Percent change of transferrin saturation | between 6 and 12 months
Percent change of hemoglobin | between 6 and 12 months

SECONDARY OUTCOMES:
Proportion of children who cleared their H. pylori infection | 45+ days after completing treatment

CONTACTS AND LOCATIONS:
Overall Officials: Victor M Cardenas, MD, MPH, PhD, Principal Investigator — University of Texas-Houston School of Public Health El Paso Regional Campus
Locations (1):
- Texas Tech University School of Medicine, El Paso, Texas, United States

REFERENCES:
- [Derived] Cardenas VM, Prieto-Jimenez CA, Mulla ZD, Rivera JO, Dominguez DC, Graham DY, Ortiz M. Helicobacter pylori eradication and change in markers of iron stores among non-iron-deficient children in El Paso, Texas: an etiologic intervention study. J Pediatr Gastroenterol Nutr. 2011 Mar;52(3):326-32. doi: 10.1097/MPG.0b013e3182054123. PMID 21336159
- [Derived] Prieto-Jimenez CA, Cardenas VM, Fischbach LA, Mulla ZD, Rivera JO, Dominguez DC, Graham DY, Ortiz M. Double-blind randomized trial of quadruple sequential Helicobacter pylori eradication therapy in asymptomatic infected children in El Paso, Texas. J Pediatr Gastroenterol Nutr. 2011 Mar;52(3):319-25. doi: 10.1097/MPG.0b013e318206870e. PMID 21336156